CLINICAL TRIAL: NCT03345459
Title: College Mental Health Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Randy P. Auerbach, Director, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002625
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Depression
Keywords: Internet-based treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomized to internet-based treatment (two-thirds of sample) or usual care (one-third of sample).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Based Treatment (ICare) (Experimental): ICare Prevent is a 7-week internet-based treatment for depression that is primarily cognitive behavior therapy but targets broad-based mechanisms related to college students.
  Interventions: Other: ICare Prevent (internet-based treatment for depression in college students)
- Usual Care (No Intervention): Participants are notified that they have elevated distress, and additionally, they are provided a list of on-campus and community resources.

INTERVENTIONS:
Other: ICare Prevent (internet-based treatment for depression in college students) — ICare Prevent (internet-based treatment for depression in college students): 7 weekly sessions and 1 booster session. Each session requires about 30-45 minutes to complete. All sessions are accessed online, and it is a guided treatment (i.e., each patient provided an eCoach).
  Arms: Internet-Based Treatment (ICare)

SUMMARY:
Depression is common and debilitating disorder which, among college students, is predictive of significant problems including higher rates of dropout and suicidal behaviors. Despite viable psychotherapeutic and pharmacological options, the majority of depressed college students, like others in the general population, do not pursue treatment. Further, barriers to care, both those involving practical issues and psychological factors, lead to high attrition rates from treatment, resulting in modest effect sizes in effectiveness trials. In reaction to these alarming figures and as a means of increasing accessibility and retention, effective internet-based treatment for depression have been developed and tested. Despite increased availability, response to internet-based treatment continues to vary substantially, yet, controlled trials show that a meaningful proportion of patients who receive internet-based therapy recover. Identifying individuals with a high likelihood of responding to internet-based treatment would enable clinicians to target this inexpensive treatment only to the patients with a high probability of responding; allowing more intensive treatments to be reserved for patients who would not respond to internet-based therapy. The development of a system to make this determination would represent a major advance and address an unmet need.

ICare is an online depression treatment that has been adapted for college students (e.g., language used, problems discussed, embedded images). Prior work by the developers of ICare have tested the internet-based treatment in diverse samples of depressed adults, and prior meta-analytic research has demonstrated that psychological treatments for depression in college students are as effective relative to trials carried out among depressed adults. The overarching goal of the study is to: (a) test whether depressed college students utilize ICare, (b) identify psychosocial and clinical characteristics that increase the likelihood of ICare utilization, and (c) identify multivariate characteristics that predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-25 years;
* Enrolled as a first year student at a participating institution;
* English fluency;
* Mild or Moderate Depression: (i) PHQ-9 score 10-14 or (ii) PHQ-9 score 15-19;
* Provide Online Consent Form.

Exclusion Criteria:

* Severe Depression: (i) PHQ-9 score ≥20;
* Endorse "3" (nearly every day) on item 9 of the PHQ-9;
* No internet access

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) administered at post-treatment | Assess depressive symptoms over the prior 2 weeks.
  Self-report questionnaire assessing depression symptoms during the past 2 weeks. Scores on the PHQ-9 range from 0-27. Lower scores are indicative of less severe depressive symptoms.
Generalized Anxiety Disorder - 7 item (GAD-7) administered at post-treatment | Assess anxious symptoms over the prior 2 weeks.
  Self-report questionnaire assessing anxiety symptoms during the past 2 weeks. Scores on the GAD-7 range from 0-21. Lower scores are indicative of less severe anxious symptoms.
EuroQol 5 (EQ-5D) administered at post-treatment | Examines problems/symptoms over the prior 2 weeks.
  Comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 items is rated on a scale from 1 to 3, and then summed to a total score. Lower scores are indicative of less severe problems.

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No